CLINICAL TRIAL: NCT00925106
Title: A Pilot, Open-Label, Randomized, Crossover, Pharmacokinetic Study Of Enhanced Bioavailability Celecoxib Formulations D1, D2 And D3 In Healthy Volunteers
Brief Title: Pharmacokinetics Of Celecoxib Test Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3191355
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
Keywords: Bioavailability, pharmacokinetics, celecoxib
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Celebrex capsule (Active Comparator): Commercial capsule
  Interventions: Drug: Celebrex capsule
- D1 (Experimental): Test formulation D1
  Interventions: Drug: Test formulation D1
- D2 (Experimental): Test formulation D2
  Interventions: Drug: Test formulation D2
- D3 (Experimental): Test formulation D3
  Interventions: Drug: Test formulation D3

INTERVENTIONS:
Drug: Celebrex capsule — Single dose 200 mg commercial Celebrex capsule
  Arms: Celebrex capsule
Drug: Test formulation D1 — Single dose 150 mg celecoxib as formulation D1
  Arms: D1
Drug: Test formulation D2 — Single dose 150 mg celecoxib as formulation D2
  Arms: D2
Drug: Test formulation D3 — Single dose 150 mg celecoxib as formulation D3
  Arms: D3

SUMMARY:
The pharmacokinetics of new formulations of celecoxib are being evaluated. They are expected to provide more favorable bioavailability characteristics than the present commercial formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers
* Body weight BMI 17.5-30.5

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease
* Positive urine drug screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
AUCinf, AUCt, Cmax | 1.5 month
Visual inspection of median plasma concentration versus time profiles resulting from each formulation | 1.5 month

SECONDARY OUTCOMES:
Tmax, half-life | 1.5 month
adverse events, laboratory tests, vital signs | 1.5 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191355&StudyName=Pharmacokinetics%20Of%20Celecoxib%20Test%20Formulations